CLINICAL TRIAL: NCT04225195
Title: An Open, Multicenter Clinical Study to Evaluate the Safety, Efficacy, and Population Pharmacokinetics of ABCD for Invasive Candidiasis and Invasive Aspergillosis
Brief Title: Amphotericin B Cholesteryl Sulfate Complex for Injection(ABCD) in the Treatment of Invasive Candidiasis and Invasive Aspergillosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC/ LXMSB201901/PRO-III/A
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Invasive Candidiasis; Invasive Aspergillosis
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amphotericin B cholesteryl sulfate complex for injection(ABCD) (Experimental): Patients with invasive candidiasis (IC) will only receive intravenous treatment with ABCD. ABCD will be administered once a day at a dose of 3-4 mg/kg.
  Patients with invasive aspergillosis (IA) will be treated with ABCD for 4 weeks first, followed by oral administration of voriconazole. ABCD dosing regimen will be the same as that for IC patients.
  Interventions: Drug: Amphotericin B cholesteryl sulfate complex for injection(ABCD)

INTERVENTIONS:
Drug: Amphotericin B cholesteryl sulfate complex for injection(ABCD) — IC patients will only receive intravenous treatment with ABCD, with the longest course of treatment up to 42 days. ABCD will be administered once a day at a dose of 3-4 mg/kg. Visit plan: screening period (D-4 to D-1), baseline period (D1), treatment period and follow-up period (14±3days after the end of the last dose of ABCD).
  IA patients will be treated with ABCD for 4 weeks first, followed by oral administration of voriconazole. The total course of treatment should be at least 6 to 12 weeks. ABCD dosing regimen will be the same as that for IC patients. Visiting plan: screening period (D-4to D-1), baseline period (D1), treatment period and follow-up period.
  Other Names: ABCD

SUMMARY:
This is an open, multicenter clinical trial of ABCD for invasive candidiasis and invasive aspergillosis.

DETAILED DESCRIPTION:
This study will evaluate the safety, efficacy and population pharmacokinetic characteristics of ABCD in the treatment of invasive candidiasis and invasive aspergillosis. About 60 patients with confirmed invasive candidiasis or confirmed/probable/possible invasive aspergillosis will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed invasive candidiasis or confirmed/probable/possible invasive aspergillosis;
2. Agree to use contraceptive measures from the date of signing the informed consent to 6 weeks after the end of the last medication;
3. Female subjects must meet one of the following conditions: surgical sterilization;menopause for at least 1 year;a negative result of serum/urine pregnancy test before enrollment.
4. Signed Informed Consent Form.

Exclusion Criteria:

1. Allergic to ABCD or azole antifungal drugs；
2. For IC patients, administration of more than 48 hours of systemic antifungal treatment within 96 hours before enrollment; or 1 dose of amphotericin B in 7 days;
3. For IA patients, administration of more than 96 hours of systemic antifungal therapy for this infection before enrollment, or 1 dose of amphotericin B in 7 days;
4. Patients with Candida endocarditis, osteomyelitis, arthritis, endophthalmitis, abscess of liver and/or spleen, suppurative thrombophlebitis, or central nervous system infection;
5. Patients with a history of drug abuse or drug dependence;
6. Chronic pulmonary aspergillosis (duration ≥ 3 months), aspergilloma or allergic bronchopulmonary aspergillosis;
7. Patients are known to have mixed invasive Candida or Aspergillus infections and/or ABCD is known to be ineffective;
8. Patients with abnormal liver function;
9. Patients with reduced renal function who require or are currently undergoing hemodialysis or peritoneal dialysis;
10. Hypokalemia, which cannot be corrected before trial treatment;
11. Expected survival time is less than 2 months;
12. Patients with cardiac function of New York Heart Association（NYHA）class III/IV;
13. Positive for HIV antibody;
14. Pregnant or lactating women;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who discontinued treatment due to study drug-related adverse events or abnormal laboratory tests, Intent-to-Treat (ITT) analysis set | 4-6 weeks
  Number of patients who discontinued treatment due to study drug-related adverse events or abnormal laboratory tests, ITT analysis set
Overall response success rate at the end of ABCD treatment, modified ITT (mITT) analysis set | 4-6 weeks
  Overall response success rate at the end of ABCD treatment, m ITT analysis set
Proportion of patients who discontinued treatment due to study drug-related adverse events or abnormal laboratory tests, ITT analysis set | 4-6 weeks
  Proportion of patients who discontinued treatment due to study drug-related adverse events or abnormal laboratory tests, ITT analysis set

SECONDARY OUTCOMES:
Overall response success rate at the end of ABCD treatment, Per Protocol Set(PPS) analysis set. | 4-6 weeks
  Overall response success rate at the end of ABCD treatment, PPS analysis set.
The proportion of patients with microbiologically effective outcome at the end of treatment, micro-mITT analysis set | 4-6 weeks
  The proportion of patients with microbiologically effective outcome at the end of treatment, micro-mITT analysis set
30-d all-cause mortality rate after starting treatment; mITT analysis set | 30 days after starting treatment
  30-d all-cause mortality rate after starting treatment; mITT analysis set

CONTACTS AND LOCATIONS:
Overall Officials: mingui wang, Principal Investigator — Huashan Hospital affiliated to Fudan University ,Shanghai, China

IPD SHARING:
Plan to Share IPD: No